CLINICAL TRIAL: NCT04337801
Title: The Effects of Acupressure on Pain After Cesarean Section: Randomized, Single-Blind, Placebo and Control Group Study
Brief Title: The Effects of Acupressure on Pain After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ilkay Arslan, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03
Record Dates: First submitted 2020-02-27; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Postpartum Women
Keywords: Acupressure; analgesia consumption; cesarean section; nursing; pain
MeSH Terms: conditions — Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: In this study, it was ensured that the women participating in the study did not know which group they were in, and thus, a one-way blinding was performed. This was performed by using closed envelope method. The participants were masked so that the women in the acupressure and placebo groups were not informed about the pressure score applied to the acupressure points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure (Experimental): The acupressure was carried out as two sessions, postpartum second (the first session of intervention) and fourth hours (the second session of intervention). The intervention was applied bilaterally and clockwise (left Pericardium 6, left Large Intestine 4, right Large Intestine 4 and right Pericardium 6) in this study. The acupressure was applied for three minutes in average, one minute for massage and two minutes for pressure per point; with an average of 12 minutes for the whole application. In addition, the pain score of the women was assessed by themselves through the VAS before the intervention (Time 1) and 15 minutes (Time 2) after the intervention at postpartum second hour. Also, it was assessed before the intervention (Time 3) and 15 minutes (Time 4) after the intervention at postpartum forth hour. Additionally, the analgesic substance and its amount applied during the application were recorded by the first researcher.
  Interventions: Other: Acupressure
- Placebo (Placebo Comparator): The Pericardium 6 and Large Intestine 4 points were slightly touched without pressure to women in the placebo group. Touches were applied to each acupressure point for three minutes similar to the acupressure group, each session of placebo lasted approximately 15 minutes. Similar to the acupressure group, In parallel with the acupressure, the pain score of the women was recorded at the postpartum second hour (Time 1) before intervention and 15 minutes later after intervention (Time 2), and at the fourth hour (Time 3) before intervention and 15 minutes later after intervention (Time 4). Additionally, the analgesic substance and its amount applied during the application were recorded by the researcher.
  Interventions: Other: Placebo
- Control Group (No Intervention): No intervention was applied to the control group except for the routine nursing care. The data collection process in the control group was conducted in parallel with the acupressure and placebo groups. Pain score of women was recorded prior to intervention in the acupressure and placebo groups. The duration of intervention in the acupressure and placebo groups was 12 minutes and the measurements were repeated 15 minutes after the intervention. The average duration between the first and the second measurements is 30 minutes in the acupressure and placebo groups. In parallel with the acupressure and placebo groups, the current pain score of the women was recorded at the postpartum second hour (Time 1) and 30 minutes later (Time 2), and at the fourth hour (Time 3) and 30 minutes later (Time 4). Additionally, the analgesic substance and its amount applied during the application were recorded by the first researcher.

INTERVENTIONS:
Other: Acupressure — The acupressure for symptom management is performed by pressing and scrubbing-like manipulations at certain points on the acupuncture meridians.
  Other Names: Placebo
  Arms: Acupressure
Other: Placebo — The placebo intervention involves touching to the Pericardium 6 and Large Intestine 4 points without pressing.
  Arms: Placebo

SUMMARY:
Purpose: To examine the effect of Pericardium 6 and Large Intestine 4 acupressure on pain and analgesia consumption in women after cesarean section.

Methods: This study was conducted in a randomized, single-blind, placebo and control group study design with 132 women, including acupressure (n=44), placebo (n=44), and control (n=44) groups. Acupressure was administered to the Pericardium 6 and Large Intestine 4 points in the second and fourth hours after cesarean section. Data were collected using the personal information form and Visual Analog Scale. This study was used the CONSORT scheme.

DETAILED DESCRIPTION:
This study was conducted in a randomized, single-blind, placebo and control group study design. The setting was a metropolitan university hospital in Turkey. The hospital had Gynecology and Obstetrics Clinics with 56 beds with 32 nurses. The study was carried out between July 2017 and July 2018 with women who voluntarily participated in the study at the second after cesarean section

A sample size was calculated using G*Power version 3. In calculating the sample size of the study, the confidence interval was determined as 95%, the power of the study was 80% and the effect size was 0.8. Based on these reference values, the sample size was determined as 114 women. However, with a 10% loss rate, the total sample size was increased to 132, comprised of the acupressure group (n=44), the placebo group (n=44), and the control group (n=44). In the data collection process, 416 women were reached.

In this study, since the parity and the type of anesthesia were the variables to be controlled, block randomization method was preferred. The version 8.2 of the Statistical Analysis System was used to determine randomization by second researcher. By creating a randomization list through the program, the multipara and primipara women and women who experienced general and spinal anesthesia were equally divided into three groups as acupressure, placebo, and control groups.

In this study, it was ensured that the women participating in the study did not know which group they were in, and thus, a one-way blinding was performed. This was performed by using closed envelope method. The participants were masked so that the women in the acupressure and placebo groups were not informed about the pressure severity applied to the acupressure points. The nurse practitioner (MA) was couldn't unmasked because of conducting the intervention in this study. Also, the statistician wasn't masked.

In the hospital where the study was conducted, women are monitored in the recovery unit for approximately one and a half hour after cesarean section. Women are then transported to the clinic. In this study, the analgesia protocol of the Akdeniz University Hospital Obstetrics and Gynecology Department was administered by the nurses to all three groups, which are acupressure, placebo, and control group. According to the analgesia protocol, in pain management after cesarean section, primarily the diclofenac sodium is administered to the women and pain score is observed. Diclofenac sodium treatment applied in the recovery unit is reported to the nurses during the transportation of the woman to the clinic. If diclofenac sodium was not administered to the women in the recovery unit, diclofenac sodium is applied through the intra muscular (IM) to them just after hospitalization following the cesarean section. Subsequent to the use of diclofenac sodium, the women are evaluated for pain score and treatment is continued with either of the analgesia among pethidine hydrochloride, diclofenac sodium, and paracetamol. Maintaining analgesia at plasma concentration is important in pain management. Maintaining analgesia in plasma concentration in women after cesarean section is performed with paracetamol.

The acupressure protocol was prepared according to previous studies, guidelines and expert opinions. Although no consensus concerning the combined points used, number of repetitions, duration, and frequency of intervention, it is recommended to combine the related points as well as using repeated sessions to increase the effect of the acupressure. In a systematic review on this subject, in the high-quality studies, compared to other points, Spleen 6 and Large Intestine 4 points were found to be more effective in managing uterine pain. In addition, in order to increase the effect of the acupressure, it is recommended to combine the related points as well as to perform repeated sessions. In this study, in order to increase the effect of the acupressure, the Pericardium 6 point (co-localization of pain and nausea-vomiting centers in the brain stem) was combined with the Large Intestine 4 point. In the postpartum period, the acupressure is applied as a manual pressure on the acupressure points to the woman lying on her back and legs straight. The acupressure was carried out by the first researcher in two sessions, postpartum second (the first session of intervention) and fourth hours (the second session of intervention). Although there was no difference in the order of use of the acupressure points, the intervention was applied bilaterally and clockwise (left Pericardium 6; left Large Intestine 4; right Large Intestine 4; and right Pericardium 6) in this study. Before the acupressure, each acupressure point was massaged for approximately a minute. Subsequently, the acupressure was applied to each point for approximately two minutes with a six second pressure and two second relaxation periods. The acupressure was applied for three minutes in average, one minute for massage and two minutes for pressure per point; with an average of 12 minutes for the whole application. In addition, the pain score of the women was assessed by themselves through the VAS before the intervention (Time 1) and 15 minutes (Time 2) after the intervention at postpartum second hour. Also, it was assessed before the intervention (Time 3) and 15 minutes (Time 4) after the intervention at postpartum forth hour. Additionally, the analgesic substance and its amount applied during the application were recorded by the first researcher.

The procedure of the placebo group was prepared in parallel with the acupressure procedure. The only difference was that the Pericardium 6 and Large Intestine 4 points were slightly touched without pressure to women in the placebo group. Touches were applied to each acupressure point for three minutes similar to the acupressure group, each session of placebo lasted approximately 15 minutes. Similar to the acupressure group, In parallel with the acupressure, the pain score of the women was recorded at the postpartum second hour (Time 1) before intervention and 15 minutes later after intervention (Time 2), and at the fourth hour (Time 3) before intervention and 15 minutes later after intervention (Time 4). Additionally, the analgesic substance and its amount applied during the application were recorded by the researcher.

No intervention was applied to the control group except for the routine nursing care. The data collection process in the control group was conducted in parallel with the acupressure and placebo groups. Pain score of women was recorded prior to intervention in the acupressure and placebo groups. The duration of intervention in the acupressure and placebo groups was 12 minutes and the measurements were repeated 15 minutes after the intervention. The average duration between the first and the second measurements is 30 minutes in the acupressure and placebo groups. In parallel with the acupressure and placebo groups, the current pain score of the women was recorded at the postpartum second hour (Time 1) and 30 minutes later (Time 2), and at the fourth hour (Time 3) and 30 minutes later (Time 4). Additionally, the analgesic substance and its amount applied during the application were recorded by the first researcher.

Data were collected by Personal Information Form and Visual Analog Scale. The version 8.2 of the Statistical Analysis System was used for statistical analysis of the data obtained from the study. Descriptive statistics of the study were evaluated with mean, Standard Deviation (SD), number, and percentage. Pearson chi-square test was used to evaluate the group homogeneity of the data. The t-test was used for comparisons between two categories of variables. In addition, variance analysis was used to find the differences among three or more categorical variables and to evaluate the data obtained at different measurement times. In the repeated measures, the paired sample t-test was used among the dependent groups for the variables that were found to be significant as a result of variance analysis. The significance level in the whole study was accepted as 0.05.

Ethics permission of the study was gained from Akdeniz University Clinical Research Ethics Committee (No: 335, Date: 31.05.2017). Participants were informed that participation in the research was voluntary, they could leave the research at any time, and the collected data will be kept completely confidential and secured. Informed consent was obtained from all individual participants included in the study.

ELIGIBILITY:
Inclusion Criteria:

* to be between 18-45 years old
* to give a birth by cesarean section between 37-40 weeks
* to give a birth to a healthy baby at the end of a singleton pregnancy
* to be in the postpartum second hour
* to have no problem that prevents verbal communication

Exclusion Criteria:

* to have the cesarean section after a high-risk pregnancy
* to have severe systemic diseases
* to have complications in the mother and/or the newborn after cesarean section
* to be administered patient controlled analgesia
* to have a body mass index over 25 kg/m2
* to have a previous acupressure experience
* to have intracath on the area of intervention
* to have smoking and alcohol use during pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
Pretest pain score in postpartum second hour | Time 1 represents the measurement time before the intervention at postpartum second hour.
  The pain score of the women was assessed by themselves through the Visual Analog Scale (VAS). The VAS is a ruler scale with a length of 10 cm, which is prepared with 1 cm intervals. On the scale, 0 stands for "no pain", 10 means "unbearable pain". In this study, the VAS was used in vertical format. Women were asked to mark their pain score on the scale.
Posttest pain score in postpartum second hour | Time 2 represents the measurement time at 15 minutes after the intervention at postpartum second hour.
  The pain score of the women was assessed by themselves through the Visual Analog Scale (VAS). The VAS is a ruler scale with a length of 10 cm, which is prepared with 1 cm intervals. On the scale, 0 stands for "no pain", 10 means "unbearable pain". In this study, the VAS was used in vertical format. Women were asked to mark their pain score on the scale.
Pretest pain score in postpartum fourth hour | Time 3 represents the measurement time before the intervention at postpartum four hour.
  The pain score of the women was assessed by themselves through the Visual Analog Scale (VAS). The VAS is a ruler scale with a length of 10 cm, which is prepared with 1 cm intervals. On the scale, 0 stands for "no pain", 10 means "unbearable pain". In this study, the VAS was used in vertical format. Women were asked to mark their pain score on the scale.
Posttest pain score in postpartum fourth hour | Time 4 represents the measurement time at 15 minutes after the intervention at postpartum fourth hour.
  The pain score of the women was assessed by themselves through the Visual Analog Scale (VAS). The VAS is a ruler scale with a length of 10 cm, which is prepared with 1 cm intervals. On the scale, 0 stands for "no pain", 10 means "unbearable pain". In this study, the VAS was used in vertical format. Women were asked to mark their pain score on the scale.

SECONDARY OUTCOMES:
Analgesic consumption before intervention at postpartum second hour | It includes the time from delivery to first intervention at the second hour of postpartum
  All women were received routine nursing care and analgesia protocol for post-cesarean pain. The analgesic consumption of women were recorded by the first researcher.
Analgesic consumption during the process after the intervention at the second hour after birth | It includes an average of 3 hour from immediately after the interventions at second hour of postpartum to study completion.
  All women were received routine nursing care and analgesia protocol for post-cesarean pain. The analgesic consumption of women were recorded by the first researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Akgün, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akgun M, Boz I. The effects of acupressure on post-cesarean pain and analgesic consumption: a randomized single-blinded placebo-controlled study. Int J Qual Health Care. 2020 Nov 16;32(9):609-617. doi: 10.1093/intqhc/mzaa107. PMID 32877509